CLINICAL TRIAL: NCT04803422
Title: Per Oral Versus Intravenous Postoperative Antibiotics After Surgery for Complicated Appendicitis: A Cluster Randomized Cluster Crossover Non-Inferiority Study.
Brief Title: Per Oral Versus Intravenous Postoperative Antibiotics After Surgery for Complicated Appendicitis.
Acronym: PIPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-2021-27
Record Dates: First submitted 2021-02-27; First posted 2021-03-17 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-07

CONDITIONS: Complicated Appendicitis
MeSH Terms: interventions — Anti-Bacterial Agents; Metronidazole; Piperacillin, Tazobactam Drug Combination; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Masking Description: An electronic randomization sequence in the program R will be applied to randomize centers (clusters) 1:1. After randomization the allocation will not be concealed
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1- Postoperative Course (Active Comparator): Pre-or intraoperative antibiotics (both uncomplicated and complicated) appendicits: Single-dose inj. Metronidazole and Pipperacillin/Tazobactam. In case of allergy to penicillin: Single-dose inj. Metronidazole and intravenous inj. Cefuroxim.
  First 6 month: Tablet Amoxicillin/Clavulanic Acid and Tablet Metronidazole.In case of allergy to Penicillin: Tablet Metronidazole and Tablet Ciprofloxacillin.
  Last 6 month: Intravenous Metronidazole and Intravenous Pipperacillin / Tazobactam. In case of allergy to penicillin: Intravenous Metronidazole and Intravenous Cefuroxim.
  Interventions: Drug: Antibiotic
- Arm 2 - Postoperative Course (Active Comparator): Pre-or intraoperative antibiotics (both uncomplicated and complicated) appendicits: Single-dose inj. Metronidazole and Pipperacillin/Tazobactam. In case of allergy to penicillin: Single-dose inj. Metronidazole and intravenous inj. Cefuroxim.
  First 6 month: Intravenous Metronidazole and Intravenous Pipperacillin / Tazobactam. In case of allergy to penicillin: Intravenous Metronidazole and Intravenous Cefuroxim.
  Last 6 month: Tablet Amoxicillin/Clavulanic Acid and Tablet Metronidazole.In case of allergy to Penicillin: Tablet Metronidazole and Tablet Ciprofloxacillin.
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Antibiotic — The study aims to test whether oral antibiotics is non-inferior compared to intravenous antibiotics.
  Other Names: metronidazole intravenous; metronidazole oral; Piperacillin / Tazobactam; Amoxicillin / Clavulanic acid

SUMMARY:
The PIPA trial is a prospective, multicentre, cluster randomized cluster crossover non-inferiority study. We aim to test whether a three-day postoperative course of per oral antibiotics is non-inferior to a three-day postoperative course of intravenous antibiotics as standard care after laparoscopic surgery for complicated appendicitis in regards to the risk of postoperative intraabdominal abscess formation within 30-days

DETAILED DESCRIPTION:
Complicated appendicitis increases the risk of postoperative intra-abdominal abscess. Treatment of complicated appendicitis are usually with a postoperative course of intravenous antibiotics. There is need for a study confirming the results of retrospective studies showing that a postoperative course of oral antibiotics is not inferior to intravenous antibiotics after laparoscopic surgery for complicated appendicitis.

The PIPA trial will be a prospective, multicenter, cluster randomized cluster crossover non-inferiority study designed to test whether a three-day postoperative course of per oral antibiotics is non-inferior to a three-day postoperative course of intravenous antibiotics as standard care after laparoscopic surgery for complicated appendicitis in regards to the risk of postoperative intraabdominal abscess formation within 30-days. Participating hospitals will be randomized to either a 6-month period with a per oral antibiotic regime followed by a 6-month period with an intravenous antibiotic regime, or 6-month period with an intravenous antibiotic regime followed by a 6-month period with a per oral antibiotic regime for the postoperative treatment after laparoscopic surgery for complicated appendicitis. Primary outcome will be the incidence of intra-abdominal abscess by the postoperative day 30.

The study duration has been extended by three months in both arms, totaling six months, due to insufficient patient recruitment. By addressing this challenge, the research team seeks to achieve a more representative sample size to ensure robust and reliable research outcomes.

ELIGIBILITY:
Inclusion Criteria:

* On cluster level, hospitals with emergency surgical admissions performing laparoscopic appendectomies are eligible for inclusion.
* On an individual level, participants are eligible for inclusion if they undergo a laparoscopic appendectomy for appendicitis (both uncomplicated and complicated), are ≥ 18 years of age, and provide a signed written consent form.

Exclusion Criteria:

* Exclusion criteria are specifically related to the therapy and individual participants will be excluded if they undergo any other procedures than laparoscopic appendectomy during index surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3193 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Intra-abdominal abscess | Assessed at postoperative day 30
  Primary outcome is defined as an imaging verified intraabdominal mass treated with drainage or antibiotics, or a surgically verified intra-abdominal abscess

SECONDARY OUTCOMES:
postoperative stay | The event is assessed at postoperative day 30. The event is determnied beginning from the time the surgery ends till the time the patient is discharged from the hospital.
  postoperative length of stay measured in hours
Complications according to Clavien-Dindo Classifcation | Assessed at postoperative day 30
  complications according to the Clavien-Dindo classification at postoperative day 30, that require in- or outpatient treatment, complications grade ≥3a according to Clavien-Dindo Classification at postoperative day 30
Costs | Assessed at postoperative day 30. Data for both in- and outpatient costs will be extracted from the Danish Health Authority
  In- and outpatient costs and overall costs of both in-and- outpatient
Wound infection | Assessed postoperative day 30
  Postoperative wound infection that require in-and - outpatient treatment. A wound infection is defined as a clinically suspected wound infection which has been treated with an opening of the wound or where antibiotics has been administered for this indication

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Slagelse Hospital, Department of Surgery, Slagelse
  - Department of Surgery, Slagelse Hospital, Slagelse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohamud AA, Zeyghami W, Kleif J, Gogenur I. Postoperative recovery in peroral versus intravenous antibiotic treatment following laparoscopic appendectomy for complicated appendicitis: a substudy of a cluster randomized cluster crossover non-inferiority study. Langenbecks Arch Surg. 2024 Oct 9;409(1):303. doi: 10.1007/s00423-024-03491-w. PMID 39379540